CLINICAL TRIAL: NCT03170986
Title: Multi-Sectoral Agricultural Intervention to Improve Nutrition, Health, and Developmental Outcomes of HIV-infected and Affected Children in Western Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Boston Children's Hospital (Other); Kenya Medical Research Institute (Other); University of California, San Francisco (Other); University of South Carolina (Other); Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); Boston University (Other)
Responsible Party: Principal Investigator, Lisa Butler, Associate Research Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H16-101UCSF
Record Dates: First submitted 2017-05-01; First posted 2017-05-31 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Child Nutrition, Child Neurobehavioral Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisectoral Agriculture and Microfinance Arm (Experimental)
  Interventions: Behavioral: Multisectoral agriculture and Microfinance Intervention
- Control Arm (No Intervention)

INTERVENTIONS:
Behavioral: Multisectoral agriculture and Microfinance Intervention
  Arms: Multisectoral Agriculture and Microfinance Arm

SUMMARY:
This study aims to test the hypothesis that a multi-sectoral agricultural and microfinance intervention designed to improve household food security, prevent antiretroviral treatment failure, and reduce co-morbidities among people living with HIV/AIDS will lead to improvements in the nutrition, health and development of children under 5 years old who reside in households of adults who participate in the Shamba Maisha intervention.

DETAILED DESCRIPTION:
HIV and AIDS has had a devastating effect on household food security and wealth in sub-Saharan Africa through the debilitation of the most productive household members, decreased household income, and increased caregiver burden. Children under five living in households affected by HIV and AIDS are at particularly high risk for food insecurity and its subsequent negative impacts on nutrition, health, and neurobehavioral development outcomes. While there is widespread agreement that interventions to reduce food insecurity and poverty may improve ongoing responses to the HIV epidemic, there is a dearth of evidence regarding the effectiveness of such interventions on the nutritional, health and neurobehavioral development outcomes of HIV-affected children. Such interventions are most needed in settings such as Nyanza Region in Western Kenya: a largely rural, agricultural area characterized by high levels of poverty, HIV, food insecurity, and child mortality.

The investigators have successfully completed a one-year pilot intervention study at two health facilities in Nyanza Region including 140 (n=72 intervention, n=68 control) HIV-infected adults on antiretroviral therapy which evaluated the potential effectiveness of an integrated, multisectoral agricultural and microfinance intervention called "Shamba Maisha" ("Farm Life"), designed to increase household food security and wealth in HIV-affected households. Shamba Maisha includes a) a microfinance loan (~$175) for purchasing agricultural implements and commodities; b) agricultural implements, purchased with the loan, including a human-powered water pump, seeds, fertilizers and pesticides; and c) education in financial management and sustainable farming practices occurring in the setting of patient support groups. The trial demonstrated the feasibility, acceptability, and short-term effectiveness of Shamba Maisha on improving household food security, diet quality and health outcomes of adults living with HIV. The investigators have also successfully completed a one-year companion pediatric study in which they tested preliminary impacts of Shamba Maisha on nutritional outcomes of HIV-affected children under 5 years old who resided in households of participants in the parent study (N=200 children and 126 primary caregivers). At baseline, the investigators observed a significant degree of undernutrition in both groups. They observed statistically significant gains in weight over time for children over six months old in the intervention group (group by time interaction, p=0.01) compared to the control group, but the sample size and follow-up time were insufficient to test effects on height. A larger sample size in a randomized design with longer follow-up period is needed for a definitive test of the effectiveness of this intervention on children's health outcomes.

The investigators now propose to leverage the infrastructure of the recently funded cluster randomized controlled trial, designed to determine the effectiveness of Shamba Maisha on HIV clinical and other health outcomes of HIV-infected adults in Western Kenya (the 'parent study'). They propose to assess the impact of the intervention on nutrition, health, and neurobehavioral development outcomes for HIV-affected children. The parent study will include 8 matched pairs of health facilities, randomized in a 1:1 ratio to the intervention and control arms, enrolling 44 HIV-infected adult participants per facility (N=704 adults, 50% female) and followed for 2 years. The proposed study will enroll and follow HIV-affected children (enrolled at age 6 to <36 months) and their primary caregiver (age >18 years) who reside in compound/homesteads of participants in the parent study (1:1 ratio, intervention and control). The study will include a minimum of 352 children (n=176 per study arm) with their primary caregiver. Specific aims are: Aim 1. To determine the effect of Shamba Maisha on nutritional, health, and neurobehavioral development outcomes of HIV-affected children under 5 years old. The investigators hypothesize that children living in intervention households will have greater somatic growth (weight-for-age, height-for-age, and weight-for-height z-scores)(primary outcome), reduced morbidity and hospitalizations, and improved neurobehavioral development outcomes (secondary outcomes) compared to children living in households that do not receive the intervention. The investigators will collect data on children's nutrition, health, and neurobehavioral development outcomes over a 2-year follow-up period. Aim 2. To understand the pathways through which Shamba Maisha may improve nutritional, health, and neurobehavioral development outcomes of HIV-affected children. The investigators hypothesize that improvements in household food security and household wealth will contribute to improved child outcomes through improvements in: child diet, caregiver physical and mental health, caregiver empowerment, and home environment pathways, and this study will provide important details about those pathways. Aim 3. To evaluate the incremental cost and cost-effectiveness of the intervention with respect to children's health outcomes (in coordination with the parent study's analysis for adults). The investigators will translate observed reduced morbidity to averted Disability Adjusted Life Years (DALYs), using disability weights from the Global Burden of Disease, estimate net costs considering the intervention and averted health care costs, and calculate incremental cost-effectiveness, as the net cost per DALY averted.

ELIGIBILITY:
Inclusion Criteria:

* Compound/homesteads are eligible to participate if it has an adult who is a participant in the parent study, Households within the compound/homesteads are eligible if it has (1) a resident related to the adult participant in the parent study, (2) >1 child(ren) 6- to 36-months old, (3) the child(ren) have a parent/primary guardian age >18 years old who resides in the compound/homestead, (4) the caregiver intends to stay in the study area for the next 24 months with the child.
* Children: Age 6- to 36-months old, resident in a household in the compound/homestead of participant in the parent study. Adults: Parent or guardian of eligible child, age >18 years old, is the primary caregiver for the child(ren), and is either a participant in parent study or resident in compound/homestead of participant in the parent study.

Exclusion Criteria:

* Households in which no resident is related to the adult participant in the parent study (e.g., non-relative renters) because unrelated household members would not be expected, in Luo society, to share human, financial, or food resources with the index participant. These situations are rare in Nyanza Region.
* Children who have severe malnutrition (below -3 z-scores of the median WHO growth standards).180 Children with severe malnutrition will be excluded because they will be referred for intensive care, including feeding support.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 704 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Weight for Length Z Score | 24 months
  Weight in KG, Length in CM

SECONDARY OUTCOMES:
Morbidity | 24 months
  Number of incident respiratory and diarrheal illnesses in prior 2 weeks
Neurobehavioral Development | 24 months
  Cognitive, Motor, and Social Development Score Using the Profile for Child Monitoring Measure

CONTACTS AND LOCATIONS:
Locations (16):
- Kenya (16):
  - Kitare, Homa Bay
  - Sindo, Homa Bay
  - Hongo Ogosa, Kisumu
  - Kisumu District Hospital, Kisumu
  - Lumumba, Kisumu
  - Nyang'Ande, Kisumu
  - Pandipieri, Kisumu
  - Railways, Kisumu
  - Minyenya, Migori
  - Muhuru Bay, Migori
  - Ngodhe, Migori
  - Nyamasare, Migori
  - Osingo, Migori
  - Oyani, Migori
  - Sori Lakeside, Migori
  - Suna Ragana, Migori

IPD SHARING:
Plan to Share IPD: No
Following publication of the main paper(s) for this study, we will make survey data publicly available in the form of an electronic database for researchers who successfully complete a registration process. Survey data will be de-identified and will not contain any direct identifiers or indirect identifiers that could identify participants by inference. Users must submit brief proposals regarding intended use of the data; the study team will determine the scientific soundness of the proposal as part of the decision for the researcher to be able to access the public use dataset.

REFERENCES:
- [Derived] Richards AL, Hiepler AJ, Frongillo EA, Khan S, Holding P, Nanga K, Kammerer B, Otieno P, Butler LM. Influence of recurrent assessments during data collection on caregivers and young children for an agricultural livelihood intervention in Kenya: a qualitative study. BMJ Open. 2024 Jun 8;14(6):e077637. doi: 10.1136/bmjopen-2023-077637. PMID 38851226

DOCUMENTS (1):
  • Informed Consent Form (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT03170986/ICF_000.pdf